CLINICAL TRIAL: NCT02354625
Title: The Safety of Autologous Human Schwann Cells (ahSC) in Subjects With Chronic Spinal Cord Injury (SCI) Receiving Rehabilitation
Brief Title: The Safety of ahSC in Chronic SCI With Rehabilitation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: W. Dalton Dietrich (Other)
Collaborators: The Miami Project to Cure Paralysis (Other)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor of Neurosurgery, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140846
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Spinal Cord Injury; Paraplegia; Quadriplegia; Tetraplegia
Keywords: Schwann cells
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ahSC transplantation (Experimental): Autologous human Schwann cells
  Interventions: Biological: Autologous human Schwann cells

INTERVENTIONS:
Biological: Autologous human Schwann cells — Schwann cells harvested from the sural nerve of the participant will be autologously transplanted into the epicenter of the participant's spinal cord injury.

SUMMARY:
The purpose of this study is to assess the safety of autologous human Schwann cell (ahSC) transplantation in participants with chronic SCI.

This trial design is phase I, open label, unblinded, non-randomized, and non-placebo controlled multiple injury cohorts.

DETAILED DESCRIPTION:
For humans with chronic SCI, we hypothesize that axons might show improved function if myelin repair is induced with the implantation of ahSC. In addition spinal cord cavitation may be reduced, and neural sprouting and plasticity may be enhanced via neurotrophic effects. In this trial, subjects will receive fitness conditioning and rehabilitation prior to transplantation in order to validate the stability of their neurological baseline and enhance their ability to undergo surgery with few complications. They will also receive fitness conditioning and rehabilitation post-transplantation to maintain health and promote neuronal activity and potential neuroplasticity.

Trial enrollment will target 2 cohorts. The first cohort will be thoracic (T) level 2-12 ASIA Impairment Scale (AIS) grade A, B, or C (n = up to 4), the second cohort will be cervical (C) level 5 through T1 AIS A, B, or C (n = up to 6). Two (2) participants with AIS grade A will be enrolled prior to enrolling a participant with AIS B or C, applicable to both cohorts.

Participants will be monitored throughout a 6 month post-transplantation evaluation period for occurrence of AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status and neurological status. Safety and efficacy assessments will be performed at weeks 1 and 2 post-transplantation and months 2 and 6 post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with traumatic SCI that occurred a minimum of 12 months prior to enrollment;
2. Between the ages of 18 and 65 at last birthday;
3. SCI between spinal levels C5-T12 as defined by the most caudal level of intact motor and sensory function on the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI);
4. ASIA Impairment Scale (AIS) grade A, B, or C at time of enrollment;
5. Lesion length less than or equal to 3 cm and lesion volume less than or equal to 2 cc, as approximated by MRI.

Exclusion Criteria:

1. Persons unable to safely undergo an MRI;
2. Persons with penetrating injury of the spinal cord or complete transection of the cord, as identified by MRI;
3. Persons with severe, uncorrected post-injury spinal deformity and/or spinal cord inadequately decompressed;
4. Persons with a cavity structure that would preclude successful transplantation, as identified by MRI;
5. Persons with syringomyelia - defined as patients with progressively enlarging cysts on T2 weighted images with associated neurological decline;
6. Persons with pre-existing conditions that would preclude satisfactory sural nerve harvest;
7. Intolerance to functional electrical stimulation of muscles;
8. Exercise induced abnormalities;
9. Range of motion of the upper or lower extremities outside functional limits for targeted fitness and rehabilitation activities;
10. Evidence of bone or joint pathology that adversely influences participation in the fitness and rehabilitation activities;
11. Fracture, dislocation, or extremity instruments (implanted or external) that adversely influences participation in the fitness and rehabilitation activities;
12. Unhealed pressure ulcer;
13. History of documented seizures, stroke, brain tumor, serious head injury, or any other intracranial problem that could increase the risk of seizures during motor evoked potentials testing;
14. Pregnant women or a positive pregnancy test in those women with reproductive potential prior to enrollment;
15. Presence of disease that might interfere with participant safety, compliance, or evaluation of the condition under study;
16. Body Mass Index (BMI) ≥ 35;
17. History of active substance abuse;
18. Persons who are current participants in any interventional trial;
19. Persons with a history of prior intrathecal or intraspinal cell therapy for SCI;
20. Persons allergic to gentamicin;
21. Persons who test positive for HIV or Hepatitis B or C virus;
22. Persons with lab values significantly outside of the upper and lower limits;
23. Persons who can independently ambulate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
International Standards of Neurological Classification of Spinal Cord Injury | Change from Baseline at 6 months
Magnetic Resonance Imaging of spinal cord | Change from Baseline at 6 months
Neuropathic Pain Symptoms Inventory | Change from Baseline at 6 months
ISCI Basic Pain dataset version2 | Change from Baseline at 6 months
Pain Diagram | Change from Baseline at 6 months
Quantitative Sensory Testing | Change from Baseline at 6 months

SECONDARY OUTCOMES:
Spinal Cord Independence Measure III | Change from Baseline at 6 months
SCI-Functional Index Computer Adaptive Testing | Change from Baseline at 6 months
10-Meter Walk Test | Change from Baseline at 6 months
2-Minute Walk Test | Change from Baseline at 6 months
Timed Up and Go | Change from Baseline at 6 months
Timed Stair Climb | Change from Baseline at 6 months
Capabilities of Upper Extremity Questionnaire | Change from Baseline at 6 months
ISCI Upper Extremity Basic dataset | Change from Baseline at 6 months
ISCI Basic Bowel dataset | Change from Baseline at 6 months
ISCI Basic Lower Urinary Tract dataset | Change from Baseline at 6 months
ISCI Basic Male and Female Sexual Function datasets | Change from Baseline at 6 months
ISCI Quality of Life dataset | Change from Baseline at 6 months
Motor Evoked Potentials | Change from Baseline at 6 months
Somatosensory Evoked Potentials | Change from Baseline at 6 months
Sympathetic Skin Response | Change from Baseline at 6 months
Graded Strength Test | Change from Baseline at 6 months
1-Repetition Maximum | Change from Baseline at 6 months
Head-up Tilt | Change from Baseline at 6 months
Guy Farrar Subject Global Impression of Change | Change from Baseline at 6 months
Modified Ashworth Scale | Change from Baseline at 6 months
Pendulum Test | Change from Baseline at 6 months
Spinal Cord Assessment Tool for Spastic reflexes | Change from Baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Levi, MD, PhD, Principal Investigator — University of Miami; James Guest, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Maher JL, Anderson KD, Gant KL, Cowan RE. Development and deployment of an at-home strength and conditioning program to support a phase I trial in persons with chronic spinal cord injury. Spinal Cord. 2021 Jan;59(1):44-54. doi: 10.1038/s41393-020-0486-7. Epub 2020 Jun 3. PMID 32493977